CLINICAL TRIAL: NCT06177678
Title: A Randomized, Open-label, Active-controlled, Phase 2a Clinical Trial to Evaluate the Efficacy and Safety of TFC-003 in Patients With Primary Open-angle Glaucoma or Ocular Hypertension
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Kukje Pharma (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KJ-TFC-007
Record Dates: First submitted 2023-12-11; First posted 2023-12-20 (Actual); Last update posted 2023-12-20 (Actual); Status verified 2023-12

CONDITIONS: Primary Open Angle Glaucoma; Ocular Hypertension
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TFC-003 (Experimental): Dorzolamide 20mg/Timolol 5mg/Brimonidine 2mg combination drug. Participants will be administered 1 drop of TFC-003 ophthalmic solution twice a day for 4 weeks.
  Interventions: Drug: TFC-003
- COSOPT ophthalmic solution (Active Comparator): Dorzolamide 20mg/Timolol 5mg combination drug. Participants will be administered 1 drop of TFC-003 ophthalmic solution twice a day for 4 weeks.
  Interventions: Drug: COSOPT ophthalmic solution

INTERVENTIONS:
Drug: TFC-003 — 1 drop of TFC-003 ophthalmic solution twice a day for 4 weeks.
  Arms: TFC-003
Drug: COSOPT ophthalmic solution — 1 drop of TFC-003 ophthalmic solution twice a day for 4 weeks.
  Arms: COSOPT ophthalmic solution

SUMMARY:
The purpose of this study was to explore the efficacy and safety of the weekly intraocular pressure change of the TFC-003 group and the dorzolamid/timolol combination group in patients with primary open-angle glaucoma or ocular hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Adult men and women over 19 years of age
* At the time of the screening visit for patients diagnosed with primary open-angle glaucoma or ocular hypertension (intraocular pressure 21 mmHg or higher), patients with a history of treatment or currently receiving treatment with 3 drugs according to the combination of domestically approved glaucoma treatment ingredients and fixed-dose combination drugs, or 2 drugs Patients whose intraocular pressure was not adequately controlled despite treatment history or current use of medications
* Those whose intraocular pressure (same eye) measured at 9 a.m.(±30min) at the randomization visit is 18 mmHg or higher and 34 mmHg or lower in one or both eyes
* For subjects with a history of intraocular pressure treatment before the randomization visit, those with a wash-out period of more than 5 times the half-life of the component with the longest half-life among the components of the treatment drug
* Those with a central corneal thickness of more than 480um and less than 600um
* Those who have heard and understood the sufficient explanation and voluntarily given written consent to participate in this clinical trial

Exclusion Criteria:

* Those with MD(mean deviation of visual field) loss of -20dB or more on visual field test
* Those who have undergone ocular laser surgery within 3 months of screening
* Those whose maximum corrected visual acuity(BCVA) is less than 0.25
* Those who have used systemic corticosteroids within 1 month of randomization
* Those who have used corticosteroids administered locally to the eye or eyelid within 2 weeks of randomization
* Those who received intraocular corticosteroids through intravitreal or sub-Tenon injection within 6 months of randomization
* Patients with chronic, recurrent or severe inflammatory eye disease
* Those who have been diagnosed and treated for an eye infection or eye inflammation other than simple conjunctivitis within 3 months of the screening visit (in the case of simple conjunctivitis, within 2 months of the screening visit)
* Persons with a history of hypersensitivity to clinical investigational drugs of their components
* Those who need to wear contact lenses on visit days and when administering clinical trial drugs
* Women and men of childbearing age who plan to become pregnant or do not intend to use medically acceptable contraception during the clinical trial periode(however, women of childbearing age who have not undergone sterilization surgery may participate in the clinical trial only if they are tested for pregnancy and the results are negative. You must agree to participate and maintain effective contraception for the entire clinical trial period).
* Currently pregnant or lactating
* Those who have suffered eye trauma or surgery within 6 months of the screening visit
* Those who are confirmed to have a positive HBsAg or HCV Ab test result at the time of screening(can be used if test results are within 6 months from the time of screening)
* Any abnormality that precludes reliable IOP measurement (e.g. corneal opacity, nystagmus, congenital cataract, damage to photosensitive tissue cells, optic neve/optic center disease/ptosis, keratoconus, etc. that precludes IOP measruement)
* Those who have a positive history of HIV Ab in the past or are confirmed to have a positive HIV Ab test result at the time of screening (can be used if the test result is within 6 months of the time of screening)
* Patients with bronchial asthma or a history of reactive airway disease, including bronchospasm and severe chronic obstructive pulmonary disease
* Patients with sinus bradycardia, 2nd or 3rd degree atrioventricular block, obvious heart failure, cardiogenic shock, sinus dysfunction syndrome, sinoatrial block
* Those taking MAO inhibitors
* People taking antidepressants that affect noradrenaline transmission (e.g. tricyclic antidepressants, mianserin)
* People with untreated pheochromocytoma
* Subjects who, in the opinion of the investigator, have other ocular pathology (severe dry eyes, etc.) that makes it impossible to administer the investigational drug
* Patients with severe renal impairment (creatinine clearance<30mL/min) or hyperchloremic acidossis
* Persons who received other investigational drugs within 30 days of randomization
* Other people deemed unsuitable for participation in this clinical trial according to the medical opinion of the investigator

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-02 (Estimated); Primary Completion 2024-09 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Average change from baseline in weekly intraocular pressure at 4 weeks | Baseline and week 4
  The Average change in intraocular pressure at 4 weeks compared to the baseline is defined as the weekly average change for measurements at 9a.m.(±30min), 11a.m.(±30min), and 2p.m.(±30min).

CONTACTS AND LOCATIONS:
Locations (1):
- Kukje Pharm, Seongnam-si, South Korea

IPD SHARING:
Plan to Share IPD: Undecided
Not yet decided.

REFERENCES:
- [Result] Kass MA, Heuer DK, Higginbotham EJ, Johnson CA, Keltner JL, Miller JP, Parrish RK 2nd, Wilson MR, Gordon MO. The Ocular Hypertension Treatment Study: a randomized trial determines that topical ocular hypotensive medication delays or prevents the onset of primary open-angle glaucoma. Arch Ophthalmol. 2002 Jun;120(6):701-13; discussion 829-30. doi: 10.1001/archopht.120.6.701. PMID 12049574
- [Result] Musch DC, Lichter PR, Guire KE, Standardi CL. The Collaborative Initial Glaucoma Treatment Study: study design, methods, and baseline characteristics of enrolled patients. Ophthalmology. 1999 Apr;106(4):653-62. doi: 10.1016/s0161-6420(99)90147-1. PMID 10201583
- [Result] Gulkilik G, Oba E, Odabasi M. Comparison of fixed combinations of dorzolamide/timolol and brimonidine/timolol in patients with primary open-angle glaucoma. Int Ophthalmol. 2011 Dec;31(6):447-51. doi: 10.1007/s10792-011-9495-z. Epub 2011 Dec 30. PMID 22207522
- [Result] Kitazawa Y, Shirai H, Go FJ. The effect of Ca2(+) -antagonist on visual field in low-tension glaucoma. Graefes Arch Clin Exp Ophthalmol. 1989;227(5):408-12. doi: 10.1007/BF02172889. PMID 2806924
- [Result] Brooks DE. Glaucoma in the dog and cat. Vet Clin North Am Small Anim Pract. 1990 May;20(3):775-97. doi: 10.1016/s0195-5616(90)50062-5. PMID 2194358
- [Result] Ishii Y, Nakamura K, Tsutsumi K, Kotegawa T, Nakano S, Nakatsuka K. Drug interaction between cimetidine and timolol ophthalmic solution: effect on heart rate and intraocular pressure in healthy Japanese volunteers. J Clin Pharmacol. 2000 Feb;40(2):193-9. doi: 10.1177/00912700022008739. PMID 10664926